CLINICAL TRIAL: NCT05331131
Title: Efficacy of Ketamine Mouthwash in the Management of Oral and Pharyngeal Toxicity
Brief Title: Efficacy of Ketamine Mouthwash in the Management of Oral and Pharyngeal Toxicity Associated With Head and Neck Chemoradiotherapy: A Phase 2, Simon 2-stage Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study team not moving forward with protocol
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-0292
Record Dates: First submitted 2022-03-24; First posted 2022-04-15 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cancer of Head and Neck; Mucositis Oral; Pharyngeal Mucositis
Keywords: Cancer of Head and Neck; Radiation Therapy; Intensity-Modulated Radiation Therapy; Concurrent chemotherapy; Ketamine; Ketamine mouthwash; Oral mucositis; Pharyngeal mucositis
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Simon 2-stage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine Mouthwash (Experimental): Enrolled patients with histologically confirmed squamous cell carcinoma of the head and neck undergoing definitive radiation therapy to 70Gy with concurrent cisplatin chemotherapy who develop grade 3+ toxicity will be prescribed ketamine mouthwash at a strength of 20mg/5mL in NovaFilm suspension with OraSweet flavoring agent via "swish and spit" route of administration. They will take the investigational drug four times daily.
  Interventions: Drug: Ketamine Topical

INTERVENTIONS:
Drug: Ketamine Topical — Ketamine hydrochloride in mouthwash form
  Other Names: Ketamine mouthwash

SUMMARY:
Patients with head and neck cancer generally receive a standard of care of 7 weeks of daily radiation therapy given alongside an aggressive chemotherapy drug called cisplatin. While rates of cure are often strong for patients who are able to complete treatment without any unscheduled breaks, the rates of high grade toxicity associated with this treatment are high even with the use of the most modern techniques of treatment. Pain, swallowing dysfunction, loss of taste sensation, and ulceration of the mouth and throat are ubiquitous and often contribute to a nutritional breakdown requiring feeding tube placement. Unfortunately, even with aggressive use of opioids and other conventional palliation methods, breakthrough pain and other toxicities are very common. In addition to the quality of life burdens of these side effects, patients who are unable to complete treatment on schedule have worse control of their cancer and worse overall survival.

Clearly, there is a clinical need for better management of these toxicities. The investigators hypothesize that ketamine mouthwash may effectively reduce both pain and the need for opioid drugs in this patient population. There is a large body of literature supporting the use of ketamine for pain control in diseases other than cancer, and a smaller but growing body of literature showing the effectiveness of ketamine for control of cancer-associated pain. Additionally, by providing ketamine in mouthwash form, the evidence shows that one can avoid the side effects associated with giving ketamine throughout the body, and in fact no significant side effects have been reported so far with this treatment.

In this study, the investigators will provide ketamine mouthwash to patients undergoing the standard treatment for this disease over a two week period, and measure their response in terms of both pain and need for opioids, as well as other measurements of quality of life. The investigators will also measure unscheduled interruptions in treatment. In years to come, the data from this study may show an impact on cancer control and survival.

DETAILED DESCRIPTION:
There is an unmet need for improvement in pain control among patients with cancer and undergoing anti-neoplastic therapies, with by one recent estimate 59% of patients on treatment and 33% of patients who completed curative treatment reporting inadequate pain control (1).

This burden is especially grave in the setting of curative treatment for head and neck cancer, in which rates of severe acute pain and other toxicities with major impact on quality of life are known to be high among radiotherapy and chemoradiotherapy patients.

In RTOG 9003, a randomized controlled trial evaluating altered fractionation in the setting of definitive radiotherapy in locally advanced head and neck cancer, acute grade 3-4 oral mucositis was seen in 25% of standard fractionation and 41% of hyperfractionation patients, and acute grade 3-4 pharyngeal/esophageal toxicity was seen in 11% of standard fractionation and 26% of hyperfractionation patients. In RTOG 0129, a randomized controlled trial evaluating accelerated fractionation in the setting of definitive cisplatin-based chemotherapy concurrent with radiotherapy in stage III-IV head and neck cancer, acute grade 3-4 dysphagia was seen in 23% of standard fractionation and 21% of accelerated fractionation patients, and acute grade 3-4 oral/pharyngeal mucositis was seen in 39% of standard fractionation and 33% of accelerated fractionation patients. Additionally, in RTOG 0129, 69% of standard and 67% of accelerated fractionation patients received nutritional support via feeding tube by treatment end (2,3).

The above landmark RTOG studies did not use modern intensity-modulated radiation therapy (IMRT) techniques which have since become standard in head and neck radiotherapy, and data do exist suggesting reduced acute toxicities through the use of IMRT such as in RTOG 0022 (4). Nevertheless, the burden is still significant, particularly when concurrent cisplatin is given. For example, in RTOG 1016, a randomized controlled trial which demonstrated the inferiority of cetuximab given concurrently with IMRT vs. concurrent cisplatin and IMRT in HPV-positive oropharyngeal cancers, the IMRT plus cisplatin arm showed an acute grade 3-4 dysphagia rate of 37.4%, an acute grade 3-4 oral mucositis rate of 41.5%, an acute grade 3-4 pharyngeal mucositis rate of 13.6%, an acute grade 3-4 anorexia rate (which is likely due at least in part to pain and swallowing dysfunction) of 22.4%, and a rate of feeding tube nutritional support at treatment end of 62% (5).

As a result of the above and other randomized studies, IMRT with concurrent cisplatin-based chemotherapy, with its high rates of expected high grade toxicities, is the standard of care for head and neck cancers except for those that are potentially operative and those that are very early stage.

Early treatment termination is common in definitive head and neck cancer treatment, and oral and pharyngeal toxicities are among the most significant factors associated with early treatment termination. In our own institution, among the 5014 new treatment starts between 2017 and 2019, curative intent head and neck cases had a 7.9% treatment termination rate, the second highest by percentage of new starts of any disease site after vulvar cancer (vs. an overall institutional rate of 4.1%), and made up 38.2% of all treatment terminations in this interval, the highest share of any disease site by far (6).

Patients who fail to complete treatment are well understood to have vastly poorer rates of control and survival than patients who do complete treatment. Additionally, head and neck patients with extended treatment package time due to unscheduled breaks have worse survival than those completing treatment on time (7,8). Therefore, therapies which can ameliorate these toxicities and thereby reduce treatment breaks, package time, and terminations, may not only improve patient quality of life but may also have a downstream beneficial impact on control and survival metrics in light of improved rates of treatment completion.

Ketamine is an anesthetic agent developed in the 1960s as a derivative of phencyclidine (PCP) to be a less toxic alternative to the latter. It maintains its position on the WHO list of essential medications and continues to see widespread use in anesthesia and is widely and inexpensively available globally. Ketamine has numerous routes of administration to fit specific clinical needs, including IV, IN, IM, SC, IT/epidural, PO, and multiple topical formulations.

Ketamine's complex pharmacology illustrates its potential benefits in the oncologic setting. Its primary mechanism of action is as a high affinity non-competitive antagonist to the NMDA receptor, driving anesthetic and analgesic effects which include decreased central sensitization to opioids. Additional mechanisms of action promoting analgesia include: reduction of extracellular D-serine with the downstream effect of reduced NMDA receptor activation; inhibition of hyperpolarization-activated cyclic nucleotide gated channels (HCNs); both potentiation and inhibition of cholinergic receptors; activation of mu-, kappa-, and delta-opioid receptors; activation of sigma receptors; inhibition of voltage gated sodium channels; reduction in activity of pro-inflammatory cytokines; and decreased astrocyte and microglial activation leading to decreased transmission of nociceptive inputs. Further therapeutic effects of ketamine include potent anti-depressant pathways, which can indirectly ameliorate pain and discomfort by altering a subject's perception of pain acuity and may also marginally improve treatment completion rates to the extent that depression is associated with treatment termination. Conversely, adverse effects of ketamine are generally transient except in the setting of heavy chronic use and are generally limited to systemic routes of administration as opposed to topical routes (9).

Clinical data support ketamine use in the oncologic setting as well. To date, five randomized controlled trials have analyzed systemic administration of ketamine to cancer patients, of which four detected either statistically significant pain reduction or reduction in opioid analgesic burden, while the fifth trial was hampered by a dose escalation design which led to study subject withdrawal due to severe psychotomimetic adverse effects (10).

Topical administration of ketamine for local pain control is a further area of active investigation. A randomized controlled trial analyzed the use of 1% ketamine cream, 2% amitriptyline cream, and combination ketamine-amitriptyline cream for control of neuropathic pain and found reductions in pain scores in all groups, although non-significantly vs. placebo. Plasma concentrations of ketamine were measured in this study and ranged from undetectable to 30ng/ml, as against a serum threshold level of 2000ng/ml for induction of psychoactive effects, indicating essentially negligible potential for systemic side effects including the feared psychotomimetic adverse effects (11,12). More broadly, a systematic review of 34 studies on topical ketamine for pain control including 13 randomized controlled trials in diverse domains including postherpetic neuralgia, diabetic neuropathy, chemotherapy-induced neuropathy, and pelvic pain found clinically and statistically significant pain reduction in the overwhelming majority of studies, with zero reported systemic side effects and maximum reported plasma levels of 33ng/ml and 20.9 ng/ml for ketamine and norketamine, respectively. Pain response to the treatment appears to be dose dependent but even at concentrations up to 20% ketamine, systemic absorption remains clinically insignificant (13).

Of particular note, topical ketamine solution has been used in two randomized controlled trials for controlling post-tonsillectomy pain in pediatric patients. One trial compared 5% ketamine administered to the tonsillar fossae with soaked swabs to a tramadol arm and a placebo, and found statistically significant improvements in pain with both interventions, with neither performing better than the other. The other trial randomized patients to 1% ketamine spray, morphine spray, lidocaine spray, or normal saline spray. Lidocaine outperformed the other groups at 20 minutes post-administration but ketamine and morphine were equally superior by 60 minutes post-administration. Neither study reported systemic or other adverse effects (14, 15).

In the oncologic setting, the NCCTG N06CA randomized controlled trial determined that a topical regimen of ketamine, baclofen, and amitriptyline for patients with chemotherapy-associated peripheral neuropathy found statistical significant improvement in motor neuropathy and a trend towards improvement in sensory neuropathy after four weeks of treatment vs. placebo, without psychoactive side effects and an overall side effect profile equivalent to placebo (16). A phase I trial of topical ketamine, amitriptyline, and lidocaine for radiation dermatitis found long-term improvement in pain and other dermatologic endpoints (17). A published case study describes a 32 year old patient with oral tongue cancer undergoing adjuvant radiation therapy to 66 Gy who had severe breakthrough pain despite aggressive interventions including transdermal fentanyl, oxycodone/acetaminophen, morphine suspension (which paradoxically exacerbated pain), "magic mouthwash," hydromorphone, and sucralfate. The patient was treated with ketamine mouthwash at a strength of 20mg/5ml, experienced significant pain relief within minutes of administration, continued regular use of ketamine mouthwash and went on to have profound and durable symptomatic improvement which additionally enabled her nutritional recovery (18).

As of this writing, one phase II trial has studied topical oropharyngeal (i.e. mouthwash) administration of ketamine in the setting of grade 3 or 4 chemotherapy-associated oral mucositis. That study found statistically significant improvements in patient-reported pain scores both at rest and when swallowing at multiple time intervals following ketamine administration, statistically significant improvement in patient reported sleep quality, and a non-statistically significant trend towards reduced median opioid analgesic burden for which the study was likely underpowered (19).

An NCT-registered randomized controlled trial is studying the analgesic efficacy of ketamine mouthwash in addition to topical anesthetics versus placebo in a population of 19 patients receiving head and neck radiation therapy or chemoradiation. This study has not yet reported results (20).

Another recently published randomized controlled trial studied the efficacy of ketamine mouthwash for chemotherapy-associated oral mucositis in the pediatric population in terms of analgesic impact and need for rescue analgesics. Only a single dose of ketamine was administered and its effects only monitored for several hours. Although differences were observed in the ketamine and placebo groups, they did not meet significance thresholds (21).

The two foregoing RCTs of ketamine mouthwash are limited by sample size, by only capturing analgesia outcomes in the former case, and by single dose administration with transient follow-up in the latter case. Nevertheless, they testify to the potential therapeutic value of ketamine mouthwash for cancer patients, and to a safety profile favorable enough for consideration its use in children.

The investigators' contention is that the above basic and clinical data, and the clear clinical need for better control of toxicity associated with anti-neoplastic therapy of head and neck cancer, justify a prospective trial investigating the use of ketamine for toxicity control in head and neck cancer patients and its attendant impact on pain control, opioid analgesic burden, functional quality of life metrics, and on-schedule completion of curative therapy as prescribed. The investigators aim to study ketamine intervention in the setting of intensity-modulated radiation therapy with concurrent cisplatin-based chemotherapy, the standard of care and most intensive current curative regimen for definitive treatment of head and neck cancer. Adjuvant therapy may also be an appropriate indication for ketamine intervention, but adjuvant cases are excluded from the present study on the grounds that post-operative recovery and complications introduce unforeseeable potential confounders in a relatively small study population.

The study agent is a mouthwash preparation of ketamine hydrochloride 20mg/5ml in NovaFilm suspension with OraSweet flavoring agent, which will be administered via swish and spit technique. Subjects will be instructed on correct administration prior to the first dose and will be observed in clinic for 1 hour following the initial administration for monitoring of AEs. Subjects will then self-administer the drug on a QID basis. They will record their self-administration (including the time of administration) in a paper drug log included among the study materials distributed to them. They will be encouraged to space administration of the drug as evenly as possible throughout the day. In order to achieve this interval of dosing, they will be encouraged to administer the drug with breakfast, lunch, dinner, and once more at bedtime. They will also be instructed that perfect uniformity of dosing schedule is not strictly necessary, and that the timing of drug administration with meals is not advised due to medical need to co-administer the drug with food, but rather to assist in adherence to the QID schedule of administration. Participants will be provided written instructions for self administration of the IP and site contact information should they have questions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-70
2. Pathologically proven squamous cell carcinoma of the oral cavity, oropharynx, nasopharynx, larynx, or hypopharynx, with the exception of stages I-II glottic cancer
3. Prescribed a curative regimen of definitive radiotherapy to with concurrent cisplatin-based chemotherapy, administered in standard fractionated doses to 70 Gy in 35 Fx
4. CTCAE v 5.0 grade 3 or greater oral cavity or pharyngeal mucositis documented to have developed subsequent to initiation of radiation therapy, defined as severe pain limiting oral intake, with at least 14 remaining days on treatment with radiation therapy

Exclusion Criteria:

1. Unable to render informed consent
2. Prior history of radiation therapy
3. Any other malignancy diagnosed or treated within 10 years prior to enrollment
4. Feeding tube placement or tracheostomy prior to initiation of radiation therapy
5. Deemed by attending radiation oncologist to be unlikely to adhere to the QID study intervention and daily outcomes reporting as described below
6. Any of the following contraindications for ketamine use: high risk for complications due to blood pressure elevation, documented hypersensitivity to ketamine, history of illicit drug use disorder, history of psychotic disorder, or any other medical contraindication attested to by the attending radiation oncologist
7. Pregnant or breastfeeding at the time of screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Assessing Pain Response | 14 days
  Pain response, defined by international consensus criteria as a combination of pain score per visual analogue scale (0-10) and opioid analgesic use (morphine-equivalent dose), through which the combination of the two measures are unified into a single evaluation of complete response (CR), partial response (PR), indeterminate response (IR), or pain progression (PP), depending upon the dynamics of VAS and MED taken separately

SECONDARY OUTCOMES:
Assessing Patient-reported pain score | Daily for 14 days
  Pain both at rest and when swallowing per Visual Analogue Scale (VAS) score from 0-10 with 10 indicating the worst pain ever felt
Measuring opioid analgesic burden | Daily for 14 days
  Total dose taken of all opioids in morphine equivalents per day on protocol
Assessing Sleep Quality | Nightly for 14 days
  Sleep quality measured by the Groningen Sleep Quality Scale from 0-14 with 14 indicating the poorest quality of sleep
Assessing Dysphagia | Baseline and repeated at 14 days
  M.D. Anderson Dysphagia Inventory with global, emotional, functional, and physical subscales of swallowing function, with a composite score from 20-100 with 100 representing maximum function
Evaluating the placement of a feeding tube | Categorical (yes/no) measurement at any time after start of ketamine therapy and prior to completion of cancer-directed therapy, a maximum 14 day period
  Feeding tube placement due to breakdown of oral intake during participation on protocol
Assessing unscheduled treatment breaks | Categorical (yes/no) measurement at any time after start of ketamine therapy and prior to completion of cancer-directed therapy, a maximum 14 day period
  Interruption at any time during participation on protocol of scheduled daily radiation fractions
Assessing premature treatment termination | Categorical (yes/no) measurement at any time after start of ketamine therapy and prior to completion of cancer-directed therapy, i.e. the time of completion of 35 fractions of radiation therapy, which may occur later than completion of the trial protocol
  Any failure to complete cancer-directed therapy as prescribed from initiation of protocol prior to final scheduled fraction of radiotherapy
Adverse events | Daily during each of the 14 days on trial protocol
  All adverse events as defined by CTCAE v. 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Bhupesh Parashar, MD, DrPH, Principal Investigator — Northwell Health
Locations (1):
- Center for Advanced Medicine, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koffler D, Eckstein J, Herman J, Martins-Welch D, Seetharamu N, Ghaly M, Kohn N, Potters L, Frank D, Sullivan K, Parashar B. Efficacy of ketamine mouthwash in the management of oral and pharyngeal toxicity associated with head and neck chemoradiotherapy: protocol for a phase II, Simon's two-stage trial. BMJ Open. 2023 Apr 11;13(4):e064809. doi: 10.1136/bmjopen-2022-064809. PMID 37041046